CLINICAL TRIAL: NCT03036839
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Ledipasvir/Sofosbuvir in Subjects With Genotype 1, 4, 5 and 6 Chronic HCV Infection Who Are on Dialysis for End Stage Renal Disease
Brief Title: Ledipasvir/Sofosbuvir in Adults With Chronic Hepatitis C Virus (HCV) Infection Who Are on Dialysis for End Stage Renal Disease
Acronym: ESRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-4063; 2016-003489-25 (EudraCT Number)
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LDV/SOF for 8 weeks (Experimental): Treatment-naive participants with genotype 1 without cirrhosis will receive LDV/SOF for 8 weeks
  Interventions: Drug: LDV/SOF
- LDV/SOF for 12 weeks (Experimental): Treatment-experienced participants with genotype 1 and treatment-naive or treatment-experienced participants with genotype 2 (Taiwan only), 4, 5 and 6 without cirrhosis will receive LDV/SOF for 12 weeks
  Interventions: Drug: LDV/SOF
- LDV/SOF for 24 weeks (Experimental): Participants with compensated cirrhosis will receive LDV/SOF for 24 weeks
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg fixed- dose combination (FDC) tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
The primary objectives of this study are to evaluate the safety, efficacy and tolerability of treatment with ledipasvir/sofosbuvir (LDV/SOF) in adults with chronic HCV infection who are on dialysis for ESRD.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic HCV infected genotype 1, 2 (Taiwan only), 4, 5, or 6 male and nonpregnant/ nonlactating females aged 18 years or older who are on dialysis for ESRD, including adults with HIV coinfection if they are suppressed on a stable, protocol-approved antiretroviral (ARV) regimens for ≥8 weeks prior to screening.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (21):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - James J. Peters VA Hospital, The Bronx, New York
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Texas Liver Institute/American Research Corporation, San Antonio, Texas
  - University of Washington/Harborview Medical Center, Seattle, Washington
- Belgium (2):
  - CUB Hopital Erasme, Brussels
  - Cliniques Universitaires UCL Saint-Luc, Brussels
- Germany (4):
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt
  - Universitatsklinikum Hamburg-Eppendorf (UKE), Zentrum fur Innere Medizin - Studienambulanz Hepatol., Hamburg
  - Ifi Studien und Projekt GmbH an der Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
- Italy (4):
  - IRCCS Ospedale Casa Sollievo Della Sofferrenza, San Giovanni Rotondo, Foggia
  - Ospedale Santa Maria Annunziata, Antella
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Background] Chuang W-L, Hu T-H, Buggisch P, et al. Ledipasvir/sofosbuvir for 8, 12, or 24 weeks is safe and effective in patients undergoing dialysis. J Hepatol 2019;70 (Suppl 1S):e225.
- [Derived] Chuang WL, Hu TH, Buggisch P, Moreno C, Su WW, Biancone L, Camargo M, Hyland R, Lu S, Kirby BJ, Dvory-Sobol H, Osinusi A, Gaggar A, Peng CY, Liu CH, Sise ME, Mangia A. Ledipasvir/Sofosbuvir for 8, 12, or 24 Weeks in Hepatitis C Patients Undergoing Dialysis for End-Stage Renal Disease. Am J Gastroenterol. 2021 Sep 1;116(9):1924-1928. doi: 10.14309/ajg.0000000000001281. PMID 34465694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Taiwan, Italy, Germany, the United States, and Belgium. The first participant was screened on 27 June 2017. The last study visit occurred on 14 February 2019.
Pre-assignment Details: 124 participants were screened.
Groups:
- LDV/SOF for 8 Weeks: Treatment-naive genotype 1 participants without cirrhosis received ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily orally with or without food for 8 weeks.
- LDV/SOF for 12 Weeks: Treatment-experienced genotype 1 participants and treatment-naive or treatment-experienced genotype 2 (Taiwan only), 4, 5, and 6 participants without cirrhosis received LDV/SOF (90/400 mg) FDC tablet once daily orally with or without food for 12 weeks.
- LDV/SOF for 24 Weeks: Participants with compensated cirrhosis received LDV/SOF (90/400 mg) FDC tablet once daily orally with or without food for 24 weeks.
Period: Overall Study
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Started | 45 | 31 | 19
Completed | 42 | 31 | 14
Not Completed | 3 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 3 | 0 | 3
Not completed — Withdrew Consent | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug. Participants were grouped within the Safety Analysis Set according to the treatment they actually received.
Groups:
- LDV/SOF for 8 Weeks: Treatment-naive genotype 1 participants without cirrhosis received LDV/SOF (90/400 mg) FDC tablet once daily orally with or without food for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks | Total
Number analyzed (Participants) | 45 | 31 | 19 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12.0) | 59 (10.1) | 65 (7.1) | 61 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 4 | 39
  Male | 29 | 12 | 15 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 45 | 31 | 17 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 21 | 29 | 11 | 61
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 3 | 0 | 2 | 5
  White | 20 | 2 | 6 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 3 | 0 | 0 | 3
  United States | 4 | 0 | 4 | 8
  Taiwan | 21 | 29 | 10 | 60
  Italy | 9 | 2 | 5 | 16
  Germany | 8 | 0 | 0 | 8
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene
  Participants
    CC | 24 | 24 | 9 | 57
    CT | 12 | 5 | 9 | 26
    TT | 9 | 2 | 1 | 12
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.8 (0.80) | 5.9 (0.95) | 5.9 (0.63) | 5.8 (0.82)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 24 | 14 | 10 | 48
  ≥ 800,000 IU/mL | 21 | 17 | 9 | 47
Cirrhosis Status [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 19 | 19
  No | 45 | 31 | 0 | 76
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 45 | 8 | 15 | 68
  Genotype 2 | 0 | 19 | 2 | 21
  Genotype 4 | 0 | 0 | 2 | 2
  Genotype 5 | 0 | 1 | 0 | 1
  Genotype 6 | 0 | 2 | 0 | 2
  Indeterminate | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment. The exact 95% confidence interval (CI) for the percentage within treatment group was based on the Clopper-Pearson method.
Time Frame: Posttreatment Week 12
Population: The Full Analysis Set (FAS) included participants who were enrolled into the study and received at least 1 dose of study drug. Participants were grouped within the Full Analysis Set by genotype and treatment group to which they were enrolled.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 45 | 31 | 19
percentage of participants | 93.3 [81.7 to 98.6] | 100.0 [88.8 to 100.0] | 84.2 [60.4 to 96.6]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Study Drug Due to an Adverse Event
Time Frame: First dose date up to Week 24
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 45 | 31 | 19
percentage of participants | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ (ie, 15 IU/mL) at 4 weeks after stopping study treatment. The exact 95% CI for the percentage within treatment group was based on the Clopper-Pearson method.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 45 | 31 | 19
percentage of participants | 97.8 [88.2 to 99.9] | 100.0 [88.8 to 100.0] | 84.2 [60.4 to 96.6]

4. Secondary Outcome: Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ (ie, 15 IU/mL) at 24 weeks after stopping study treatment. The exact 95% CI for the percentage within treatment group was based on the Clopper-Pearson method.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 45 | 31 | 19
percentage of participants | 93.3 [81.7 to 98.6] | 100.0 [88.8 to 100.0] | 84.2 [60.4 to 96.6]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Description: The total number of participants with HCV RNA < LLOQ was the sum of the number of participants with HCV RNA "< LLOQ detected" plus the number of participants with HCV RNA "< LLOQ target not detected (TND)". LLOQ was 15 IU/mL. The exact 95% CI for the percentage within treatment group was based on the Clopper-Pearson method.
Time Frame: Weeks 2, 4, 6, 8, 12, 16, 20, 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 45 | 31 | 19
percentage of participants
  Week 2 | 84.4 [70.5 to 93.5] | 90.3 [74.2 to 98.0] | 84.2 [60.4 to 96.6]
  Week 4: number analyzed (Participants) | 44 | 31 | 19
  Week 4 | 100.0 [92.0 to 100.0] | 100.0 [88.8 to 100.0] | 100.0 [82.4 to 100.0]
  Week 6: number analyzed (Participants) | 44 | 31 | 19
  Week 6 | 100.0 [92.0 to 100.0] | 100.0 [88.8 to 100.0] | 94.7 [74.0 to 99.9]
  Week 8: number analyzed (Participants) | 44 | 31 | 18
  Week 8 | 100.0 [92.0 to 100.0] | 100.0 [88.8 to 100.0] | 100.0 [81.5 to 100.0]
  Week 12: number analyzed (Participants) | 0 | 31 | 17
  Week 12 |  | 100.0 [88.8 to 100.0] | 100.0 [80.5 to 100.0]
  Week 16: number analyzed (Participants) | 0 | 0 | 17
  Week 16 |  |  | 100.0 [80.5 to 100.0]
  Week 20: number analyzed (Participants) | 0 | 0 | 17
  Week 20 |  |  | 100.0 [80.5 to 100.0]
  Week 24: number analyzed (Participants) | 0 | 0 | 16
  Week 24 |  |  | 100.0 [79.4 to 100.0]

6. Secondary Outcome: HCV RNA
Time Frame: Weeks 2, 4, 6, 8, 12, 16, 20, 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 44 | 31 | 19
log10 IU/mL
  Week 2: number analyzed (Participants) | 42 | 31 | 19
  Week 2 | 1.17 (0.107) | 1.22 (0.261) | 1.18 (0.098)
  Week 4 | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Week 6: number analyzed (Participants) | 44 | 31 | 18
  Week 6 | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Week 8: number analyzed (Participants) | 44 | 31 | 18
  Week 8 | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Week 12: number analyzed (Participants) | 0 | 31 | 17
  Week 12 |  | 1.15 (0.000) | 1.15 (0.000)
  Week 16: number analyzed (Participants) | 0 | 0 | 17
  Week 16 |  |  | 1.15 (0.000)
  Week 20: number analyzed (Participants) | 0 | 0 | 17
  Week 20 |  |  | 1.15 (0.000)
  Week 24: number analyzed (Participants) | 0 | 0 | 16
  Week 24 |  |  | 1.15 (0.000)

7. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Weeks 2, 4, 6, 8, 12, 16, 20, 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 44 | 31 | 19
log10 IU/mL
  Change at Week 2: number analyzed (Participants) | 42 | 31 | 19
  Change at Week 2 | -4.63 (0.799) | -4.71 (0.894) | -4.67 (0.631)
  Change at Week 4 | -4.61 (0.805) | -4.79 (0.950) | -4.71 (0.631)
  Change at Week 6: number analyzed (Participants) | 44 | 31 | 18
  Change at Week 6 | -4.61 (0.805) | -4.79 (0.950) | -4.81 (0.474)
  Change at Week 8: number analyzed (Participants) | 44 | 31 | 18
  Change at Week 8 | -4.61 (0.805) | -4.79 (0.950) | -4.81 (0.474)
  Change at Week 12: number analyzed (Participants) | 0 | 31 | 17
  Change at Week 12 |  | -4.79 (0.950) | -4.79 (0.480)
  Change at Week 16: number analyzed (Participants) | 0 | 0 | 17
  Change at Week 16 |  |  | -4.79 (0.480)
  Change at Week 20: number analyzed (Participants) | 0 | 0 | 17
  Change at Week 20 |  |  | -4.79 (0.480)
  Change at Week 24: number analyzed (Participants) | 0 | 0 | 16
  Change at Week 24 |  |  | -4.75 (0.466)

8. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Baseline up to Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 45 | 31 | 19
percentage of participants | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants Who Developed Resistance to LDV and SOF
Time Frame: Baseline up to Posttreatment Week 24
Population: The Resistance Analysis Population was defined as all participants in the Safety Analysis Set with a virologic outcome and at least 1 gene sequenced. As no participant had a relapse in this study, this outcome could not be analyzed.
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Pharmacokinetics (PK) Parameter: AUCtau of LDV
Description: AUCtau is defined as the population PK derived area under the concentration versus time curve of the drug over the dosing interval.
Time Frame: Sparse PK Samples at Weeks 6, 8, and 12 (all participants). Intensive PK samples at predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose once at Weeks 6, 8, or 12 (participants who enrolled in the optional PK substudy (N=2))
Population: The PK Analysis Set included all participants who took at least 1 dose of the study drug and had at least 1 nonmissing postdose concentration value for the corresponding analyte in plasma.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 44 | 31 | 19
h*ng/mL | 11923.9 (6319.41) | 13632.7 (4648.74) | 13542.5 (6322.88)

11. Secondary Outcome: PK Parameter: AUCtau of SOF
Description: as for outcome 10
Time Frame: as for outcome 10
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 24 | 23 | 12
h*ng/mL | 2435.4 (452.83) | 2296.6 (583.30) | 2838.2 (438.93)

12. Secondary Outcome: PK Parameter: AUCtau of GS-331007 (Metabolite of SOF)
Description: as for outcome 10
Time Frame: as for outcome 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 44 | 31 | 19
h*ng/mL | 234980.1 (67648.52) | 269050.3 (93600.65) | 280829.5 (93618.16)

13. Secondary Outcome: PK Parameter: Cmax of LDV
Description: Cmax is defined as the population PK derived maximum concentration of the drug.
Time Frame: as for outcome 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 44 | 31 | 19
ng/mL | 544.2 (271.72) | 618.4 (204.87) | 607.0 (267.38)

14. Secondary Outcome: PK Parameter: Cmax of SOF
Description: Cmax is defined as the population PK derived maximum concentration of the drug.
Time Frame: as for outcome 10
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 24 | 23 | 12
ng/mL | 1059.8 (251.74) | 1005.8 (204.54) | 1052.5 (295.06)

15. Secondary Outcome: PK Parameter: Cmax of GS-331007 (Metabolite of SOF)
Description: Cmax is defined as the population PK derived maximum concentration of the drug.
Time Frame: as for outcome 10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
Number analyzed (Participants) | 44 | 31 | 19
ng/mL | 9956.3 (2846.07) | 11392.7 (3938.33) | 11882.4 (3951.04)

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to Week 24 plus 30 days; All-Cause Mortality: First dose date up to Posttreatment Week 24
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug. Participants were grouped within the Safety Analysis Set according to the treatment they actually received.
Arm/Group | LDV/SOF for 8 Weeks | LDV/SOF for 12 Weeks | LDV/SOF for 24 Weeks
All-Cause Mortality (participants affected / at risk) | 3/45 | 0/31 | 3/19
Serious Adverse Events (participants affected / at risk) | 4/45 | 2/31 | 6/19
Other Adverse Events (participants affected / at risk) | 23/45 | 28/31 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF for 8 Weeks (N=45) | LDV/SOF for 12 Weeks (N=31) | LDV/SOF for 24 Weeks (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF for 8 Weeks (N=45) | LDV/SOF for 12 Weeks (N=31) | LDV/SOF for 24 Weeks (N=19)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 4
Chest discomfort (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 3 | 2 | 2
Influenza like illness (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 1
Tenderness (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 7 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Shunt infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 3 | 0 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 7 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 4 | 1
Headache (Nervous system disorders) | 3 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03036839/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT03036839/SAP_001.pdf